CLINICAL TRIAL: NCT04439305
Title: MATCH Treatment Subprotocol X: Phase II Study of Dasatinib in Patients With Tumors With DDR2 Mutations
Brief Title: Testing Dasatinib as a Potential Targeted Treatment in Cancers With DDR2 Genetic Changes (MATCH-Subprotocol X)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: zero accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-03342; NCI-2020-03342 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-X (Other: ECOG-ACRIN Cancer Research Group); EAY131-X (Other: CTEP); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-06

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Multiple Myeloma | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (dasatinib) (Experimental): Patients receive dasatinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Dasatinib Hydrate; Dasatinib Monohydrate; Sprycel

SUMMARY:
This phase II MATCH treatment trial identifies the effects of dasatinib in patients whose cancer has a genetic change called DDR2 mutation. Dasatinib may block proteins called tyrosine kinases, which may be needed for cancer cell growth. Researchers hope to learn if dasatinib will shrink this type of cancer or stop its growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive dasatinib orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months if less than 2 years from study entry, and then every 6 months for year 3 from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol prior to registration to treatment subprotocol
* Patients must have one of the following missense mutations in DDR2: S768R, I638F, L239R
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)
* Patients with known left ventricular dysfunction must have an echocardiogram (ECHO) or a nuclear study (multigated acquisition scan [MUGA] or First Pass) within 4 weeks prior to registration to treatment and must not have left ventricular ejection fraction (LVEF) < institutional lower limit of normal (LLN). If the LLN is not defined at a site, the LVEF must be > 50% for the patient to be eligible

Exclusion Criteria:

* Patients must not have known hypersensitivity to dasatinib or compounds of similar chemical or biologic composition
* Patients with prior use of dasatinib will be excluded
* Dasatinib should NOT be given in the presence of STRONG CYP 3A4 inhibitors/inducers. Patients who take these drugs concurrently are ineligible for treatment with dasatinib. These drugs must be discontinued prior to initiation of dasatinib
* Dasatinib should NOT be given in the presence of H2-antagonists or proton pump inhibitors. Patients who take these drugs concurrently are ineligible for treatment with dasatinib. These drugs must be discontinued prior to initiation of dasatinib. Antacids taken 2 hours before or after dasatinib administration can be used in place of H2-antagonists or proton pump inhibitors if some acid-reducing therapy is needed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2018-06-07 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Tumor assessments occurred at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
  ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among eligible and treated patients. Objective response rate is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. For each treatment arm, 90% two-sided binomial exact confidence interval will be calculated for ORR.

SECONDARY OUTCOMES:
Overall survival (OS) | Assessed every 3 months for =< 2 years and every 6 months for year 3
  OS is defined as time from treatment start date to date of death from any cause. Patients alive at the time of analysis are censored at last contact date. OS will be evaluated specifically for each drug (or step) using the Kaplan-Meier method.
Progression free survival (PFS) | Assessed at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
  Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. PFS will be estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Mary D Chamberlin, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States